CLINICAL TRIAL: NCT05410171
Title: Machine Learning-based Early Clinical Warning of High-risk Patients
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Southeast University, China (Other)
Responsible Party: Principal Investigator, Songqiao Liu, Head of Information Division, Southeast University, China
Allocation: Non-Randomized | Model: Sequential | Masking: None | Purpose: Health Services Research
Other Study IDs: 2021ZDSYLL346-P01
Record Dates: First submitted 2022-06-04; First posted 2022-06-08 (Actual); Last update posted 2022-12-01 (Actual); Status verified 2022-11

CONDITIONS: High-risk Patients; Risk Reduction; Machine Learning
MeSH Terms: conditions — Risk Reduction Behavior

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- AI group (Experimental): patients evaluated by early warning platform
  Interventions: Device: early warning platform
- usual care group (No Intervention): patients not evaluated by early warning platform

INTERVENTIONS:
Device: early warning platform — High risk inpatients will be evaluated by early warning platform
  Arms: AI group

SUMMARY:
Through the early warning platform for inpatients established by our hospital, the various indicators of patients collected in real time are carried out for automated intelligent evaluation and analysis, early warning of high-risk patients to assess the impact on patient prognosis and the impact on the occurrence of adverse events in inpatients.

DETAILED DESCRIPTION:
Build the early warning system.

ELIGIBILITY:
Inclusion Criteria:

1. Patients who use ECG monitoring
2. Age ≥ 18 years old
3. Understand and sign an informed consent form

Exclusion Criteria:

* Pregnancy or lactation

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1000 (Estimated)
Dates: Start 2022-06-01 (Actual); Primary Completion 2023-06-01 (Estimated); Study Completion 2023-12-01 (Estimated)

PRIMARY OUTCOMES:
28-day all cause mortality | 28 days
  28-day all cause mortality

SECONDARY OUTCOMES:
Hospital mortality | through study completion, an average of 1 month
  Hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Songqiao Liu, PhD., Principal Investigator — Zhongda Hospital, Southeast University, China
Locations (1):
- Zhongda Hospital, Southeast University, Nanjing, Jiangsu, China